CLINICAL TRIAL: NCT03787459
Title: Oseltamivir and Arbidol Combination Antiviral Therapy Versus Oseltamivir Monotherapy for the Treatment of Severe inﬂuenza: a Multicentre, Double-blind, Randomised Phase 3 Trial
Brief Title: Severe Influenza Trial of ARbidol
Acronym: STAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: University of Oxford (Other); Peking University (Other); National Institute for Viral Disease Control and Prevention, Chinese Center for Disease Control and Prevention (Other Government)
Responsible Party: Principal Investigator, Bin Cao, China-Japan Friendship Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAP-China Arbidol
Record Dates: First submitted 2018-12-22; First posted 2018-12-26 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-01

CONDITIONS: Influenza
Keywords: severe influenza, arbidol, oseltamivir, ordinal scale
MeSH Terms: conditions — Influenza, Human | interventions — umifenovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oseltamivir plus placebo (Active Comparator)
  Interventions: Drug: Placebos
- oseltamivir plus arbidol (Experimental)
  Interventions: Drug: Arbidol

INTERVENTIONS:
Drug: Arbidol — Oseltamivir plus Arbidol will be administrated from Days 1-7.
  Arms: oseltamivir plus arbidol
Drug: Placebos — Oseltamivir plus placebos will be administrated from Days 1-7.
  Arms: oseltamivir plus placebo

SUMMARY:
This is a multicenter, randomised, double-blind, controlled study to assess the efficacy and safety of arbidol plus oseltamivir, compared with oseltamivir alone in approximately 200 hospitalized adults and adolescent patients with confirmed severe influenza. Patients should be randomised as soon as possible after screening (no later than 12 hours), providing they are within 7 days of symptom onset. Patients will be assigned in a 1:1 ratio to receive an arbidol plus oseltamivir, or oseltamivir plus placebo. Rescreening of patients who fail to meet the inclusion and exclusion criteria will be permitted only once, providing the time from symptom onset to randomization is still within 7 days.

Arbidol/placebo will be administrated as 200mg TID from Days 1-7. Oseltamivir will be administered as 75mg twice daily from Days 1-7 (dose to be adjusted for renal impairment). Oseltamivir could be continued till influenza PCR negative. Both drugs, along with the corresponding placebo for arbidol, will be started at the time of randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized males or females with a positive antigen or PCR test for influenza virus infection
2. Age ≥16 years at the time of signing Informed Consent Form
3. Arterial oxygen saturation (SaO2)/ pulse oxygen saturation (SPO2) ≤94% in room air condition
4. ≤ 7 days since symptom onset. The onset of symptoms is defined as either: Time of the first increase in body temperature (an increase of at least 1ºC from normal body temperature- ≥38℃); Time when the patient experiences at least one general or respiratory symptom.
5. Willingness to use contraception for 7 days after the end of treatment

Exclusion Criteria:

1. Physicians make a decision that trial involvement is not in patients' best interest, or any condition that does not allow the protocol to be followed safely.
2. Patient refusal to accept invasive organ support treatment if needed
3. More than 3 consecutive doses of NAIs within 2 days before enrolment (including oseltamivir, zanamivir, peramivir)
4. Women who are pregnant (including a positive pregnancy test at enrolment), breastfeeding, or within 2 weeks post-partum.

   The following female subjects do not need to undergo a pregnancy test at enrolment: a. Postmenopausal (defined as cessation of regular menstrual periods for 2 years or more and confirmed by a follicle-stimulating hormone test) women. b. Women who are surgically sterile by hysterectomy, bilateral oophorectomy, or tubal ligation.
5. Any condition requiring renal replacement therapy
6. Severe liver disease (Child-Pugh score ≥ C)
7. A history of hypersensitivity to arbidol or oseltamivir (Tamiflu®)
8. Currently or have been involved in another anti-influenza treatment trial in the last 28 days
9. Patients who, in the opinion of the investigator, would be unlikely to comply with required study visits, self-assessments, and interventions

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2023-04-09 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint was time to clinical status improvement (the event) up to 28 days | 28 days
  the event defined as seven-category ordinal scale of clinical status after enrolment decrease by two category or discharged

SECONDARY OUTCOMES:
Time to decline of one category on the seven-category ordinal scale of clinical status lasting for 48h, or hospital discharge within 28 days, days | Up to 28 days
  the event defined as seven-category ordinal scale of clinical status after enrolment decrease by one category or discharged
Day 28 mortality rate | 28 days
Proportion of Clinical Improvement (≥2-category decline / discharge with improvement) at Days 7, 14, and 28 since arbidol initiation | Up to 28 days
Proportion of Patients at Each Category of the 7-category Ordinal Scale at Days 7, 14, and 28 | up to 28 days
Duration of Mechanical Ventilation (days), Oxygen Therapy (days), Hospitalization (days), Time from Randomization to Discharge (days), Time from Randomization to Death (days) | Up to 28 days
Incidence of Secondary Infection, Secondary Aspergillus and Bacterial Infection | Up to 28 days
Patients Requiring Continuous Renal Replacement Therapy (CRRT) After Treatment | Up to 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Dear Sir/Madam Our study receives a grant from China Ministry of Science and Technology. We cannot decide whether the data could be shared. Hope you can understand.
  Best